CLINICAL TRIAL: NCT05582187
Title: A Phase 1, Open-label, Single-dose, Parallel Cohort Study to Assess the Pharmacokinetics and Safety of Fosmanogepix (PF 07842805) in Adult Participants With Varying Degrees of Hepatic Impairment
Brief Title: A Clinical Trial of the Study Medicine (Called Fosmanogepix) in Participants With Varying Degrees of Hepatic Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4791019
Expanded Access: NCT06433128 (Available)
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Impairment
Keywords: fosmanogepix; manogepix; hepatic impairment; PF-07842805; APX001; APX001a

STUDY DESIGN:
Intervention Model Description: This is an open label, single dose, parallel cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Fosmanogepix participants with mild hepatic impairment (Experimental): Participants with mild hepatic impairment will receive a single dose of fosmanogepix, administered orally as 1 fosmanogepix tablet under fasted conditions.
  Interventions: Drug: Fosmanogepix
- Cohort 2: Fosmanogepix Participants with moderate hepatic impairment (Experimental): Participants with moderate hepatic impairment will receive a single dose of fosmanogepix, administered orally as 1 fosmanogepix tablet under fasted conditions.
  Interventions: Drug: Fosmanogepix
- Cohort 3: Fosmanogepix Participants with severe hepatic impairment (Experimental): Participants with severe hepatic impairment will receive a single dose of fosmanogepix, administered orally as 1 fosmanogepix tablet under fasted conditions.
  Interventions: Drug: Fosmanogepix
- Cohort 4: Fosmanogepix Participants with normal hepatic function (control group) (Experimental): Participants with normal hepatic function will receive a single dose of fosmanogepix, administered orally as 1 fosmanogepix tablet under fasted conditions.
  Interventions: Drug: Fosmanogepix
- Cohort 5: Fosmanogepix Participants with severe hepatic impairment (new dose level) (Experimental): Participants with severe hepatic impairment will receive a single dose of fosmanogepix, administered orally as 2 fosmanogepix tablets under fasted conditions.
  Interventions: Drug: Fosmanogepix

INTERVENTIONS:
Drug: Fosmanogepix — a single dose of fosmanogepix administered by mouth under fasted conditions

SUMMARY:
The primary purpose of this open-label study is to characterize the plasma pharmacokinetics (PK) of manogepix (active moiety of fosmanogepix) in participants with varying degrees of hepatic function following administration of a single oral dose of fosmanogepix.

All participants will receive 1 dose of fosmanogepix by mouth before breakfast on the first day at the study clinic. Serial blood samples will be collected to understand how fosmanogepix is changed and eliminated from the body. Participants will also receive physical examination and other tests. This will help to understand if fosmanogepix is safe.

Participants will be involved in this study for 4 to 9 weeks (maximum). There will be 2 to 4 study visits at the study clinic.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 17.5 to 40.0 kg/m2 (42 kg/m2 for participants of Cohort 3), inclusive; and a total body weight greater than 50 kg (greater than 110 lb)
* For participants with hepatic impairment (Cohorts 1-3, and Cohort 5): Stable hepatic impairment that meets the criteria for Class A, B, or C of the Child Pugh classification with no clinically significant change in disease status within the 28 days prior to the screening visit
* For participants with normal hepatic function (Cohort 4): No clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests
* Stable concomitant medications for the management of individual participants' medical history

Key Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection);
* Ongoing medical history of neurological disorders including abnormal movements or seizures (Note exception: stable history of peripheral neuropathy);
* Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy;
* A diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography scan, or MRI;
* Signs of clinically active Grade 2, 3 or 4 hepatic encephalopathy (ie, equal or greater than Grade 2 Portal Systemic Encephalopathy score)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose
Unbound Maximum Observed Plasma Concentration (Cmaxu) of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose
Unbound Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClastu) of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose
Unbound Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)u] of manogepix | pre-dose, 1, 2, 3, 4, 5, 6, 12, 24, 48, 96, 168, 240 hours postdose

SECONDARY OUTCOMES:
Number of Participants Reporting Treatment-emergent adverse events (AEs) | Screening to follow-up (Day 28-35)
Number of participants with clinically significant change from baseline in vital signs | From Day -1 to Day 11
Number of participants with clinically significant change from baseline in laboratory parameters | From Day -1 to Day 11
Number of participants with clinically significant change from baseline in electrocardiogram (ECG) findings | From Day -1 to Day 11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Inland Empire Liver Foundation, Rialto, California
  - Genesis Clinical Research, LLC, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT05582187/ICF_000.pdf